CLINICAL TRIAL: NCT04167215
Title: Aesthetic Analysis of Gluteal Deformity After Weight Loss and Assessment the Role of Autologous Tissue Augmentation for Gluteal Contouring
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Kamal Kamel, Teaching assistant plastic surgery departement, Assiut University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: body contouring
Record Dates: First submitted 2019-11-09; First posted 2019-11-18 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Body Contouring

STUDY DESIGN:
Intervention Model Description: assessment the role of autologous augmentation in management of different buttock deformity by using either perforator flaps or fat injection
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- perforator flap augmentation (Experimental): Doppler probe is used to locate perforating vessels from the superior gluteal artery. . Flaps or lumbar artery flap will be designed to allow deepithelialization and dissection laterally to medially to identify the perforator . then sketolization is performed A gluteal pocket will then create for the augmentation flaps by undermining in a plane just superficial to the gluteal muscle extending to within 5 cm of the inferior gluteal crease. The deepithelialized flaps will then transpose inferomedially , and tacked to the fascia with several sutures.to be used as autologus buttock augmentation flap
  Interventions: Procedure: superior gluteal artery flap and lumbar artery falp; Procedure: The gluteal pocket; Procedure: infragluteal dermal lifiting flap
- fat injection (Experimental): liposuction is performed firstly to parts where excess fat is exist and we will prepare the aspirated fat for injection as a graft in subcutaneous tissue of the buttock regoin
  Interventions: Procedure: superior gluteal artery flap and lumbar artery falp; Procedure: The gluteal pocket; Procedure: infragluteal dermal lifiting flap

INTERVENTIONS:
Procedure: superior gluteal artery flap and lumbar artery falp — Doppler ultrasound will be used to confirm location of the superior gluteal artery perforators or lumbar perforators . Flaps will be designed to allow deepithelialization and dissection . After complete sketolization of the flap it will be analyzed for viability and trimmed to achieve the desired bulk.
Procedure: The gluteal pocket — pocket will be created by undermining in a plane just superficial to the gluteal muscle from the lower body lift line inferiorly extending to within 5 cm of the inferior gluteal crease. should extend only over the medial half of the buttock.
Procedure: infragluteal dermal lifiting flap — dermal flap will be performed for lifting the ptotic buttocks with ill-defined infragluteal fold. This deepithelialized dermal flap allows for the creation of a well-defined stable infragluteal fold through an incision of the infragluteal fold and exposure of ischial tuberosity and anchor it to the ischial tuberosity.

SUMMARY:
this study aim to evaluate the role of autologous augmentation for buttock contouring and analyze different aethetic gluteal deformity

DETAILED DESCRIPTION:
The last decades showed an increasing demand for bariatric surgery and diet dependent massive weight loss , these successful strategies for weight loss result in significant deformities in general body contour , buttock normal appearance is very important for posterior trunk aesthetic image and its severely affected after massive weight loss .

Aesthetically attractive buttocks required special features include adequate volume, projection, and a defined infragluteal fold.. The gluteal region in patients with massive weight loss is characterized by excessive skin and exaggerated fat loss. Lower body lift procedures remove excess skin and lift sagging buttock tissue. unsatisfactory buttock shape especially V shaped buttock is considered as important indication for gluteal reshaping Mendieta and Cuenca-Guerra and Quezada have proposed novel methods of describing and analyzing gluteal aesthetics.

There are a multitude of options that can be used to improve the buttock includ-ing non-surgical injections, implants, fat, excisional, liposuction and various energy devices

ELIGIBILITY:
Inclusion Criteria:

* Female patients.
* patients who are seeking for gluteal contouring after massive weight loss
* age above 18 years and fixed weight for 6months.

Exclusion Criteria:

* Male patients
* Patients that will refuse the procedure,
* patients who thad a residual body mass index greater than 35
* patients have uncontrolled medical conditions.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Analysis of different gluteal deformity as regarding gluteal projection ptosis and waist hip ratio. | 2 years
  Analysis of gluteal projection will be performed using Gonzalez-ulloa method , four points and two distances , (A) Greater trochanter, (B) Point of maximal projection of the mons , (C) Point of maximal gluteal projection, (D) Anterior superior iliac spine. The CB line points to the maximal ideal projection of the buttocks. The ideal proportion is a 2:1 ratio between AB and AC.
Analysis of gluteal deformity after massive weight loss regarding gluteal ptosis | 2 years
  buttock ptosis: Gonzalez system will be used for analysis Through two lines one crossing the ischial tuber, "T" line, other crossing the mid thigh "M" lin.degrees from 0 to 7 degrees according to the definition of the crease from T to M line and the ptotic tissue surpasses the gluteal crease caudally in centimeters .
Analysis of gluteal deformity after massive weight loss regarding waist hip ratio. | 2 years
  Waist hip ratio assessment The ideal female figure has a waist-to-hip ratio of 0.7. The ration is measured in posterior view and in lateral view with the most pleasing ratio 0.65 and 0.7 respectively.
  WHO recommendation for WHR measure ; while patient being in the standing position parallel to the floor at the level at which the measurement is made and using a stretch-resistant tape and placement of the tape The measurement should be taken around the widest portion of the buttocks. at two definite point for the waist and the hip .
  For waist circumference:
  The measurement is made at the approximate midpoint between the lower margin of the last palpable rib and the top of the iliac crest.
  For hip circumference:
  The measurement should be taken around the widest portion of the buttocks.
Assessment the role of autologous flaps for gluteal contouring. | 2 years
  aesthetic analysis of the cases is described using photography and contour measures to outline the effect of the autologous flap in contour correction .
  In addition to complete review of perioperative and postoperative complications will be documented.
patient satisfaction from surgery . | 2 years
  Patients will be asked to rate the improvement of the appearance of the buttock area and their overall satisfaction with that aspect of the surgery on a 1 (no improvement) to 5 (extremely satisfied) scale
surgery complications. | 2 years
  complete review of perioperative and postoperative complications will be documented.

REFERENCES:
- [Background] Richter DF, Stoff A. Circumferential body contouring: the lower body lift. Clin Plast Surg. 2014 Oct;41(4):775-88. doi: 10.1016/j.cps.2014.07.004. PMID 25283462
- [Background] Colwell AS, Borud LJ. Autologous gluteal augmentation after massive weight loss: aesthetic analysis and role of the superior gluteal artery perforator flap. Plast Reconstr Surg. 2007 Jan;119(1):345-356. doi: 10.1097/01.prs.0000244906.48448.5d. PMID 17255692
- [Background] Centeno RF. Gluteal aesthetic unit classification: a tool to improve outcomes in body contouring. Aesthet Surg J. 2006 Mar-Apr;26(2):200-8. doi: 10.1016/j.asj.2006.01.001. PMID 19338900
- [Background] Pascal JF, Le Louarn C. Remodeling bodylift with high lateral tension. Aesthetic Plast Surg. 2002 May-Jun;26(3):223-30. doi: 10.1007/s00266-002-1478-z. PMID 12140705
- [Background] Gonzalez-Ulloa M. Torsoplasty. Aesthetic Plast Surg. 1979 Dec;3(1):357-68. doi: 10.1007/BF01577875. PMID 24174007
- [Background] Offman SL, Geddes CR, Tang M, Morris SF. The vascular basis of perforator flaps based on the source arteries of the lateral lumbar region. Plast Reconstr Surg. 2005 May;115(6):1651-9. doi: 10.1097/01.prs.0000161464.11134.c1. PMID 15861070